CLINICAL TRIAL: NCT07363746
Title: Implementation and Evaluation of a Novel Pain School Intervention Targeting Patients With Chronic Non-cancer Pain as a Tool to Achieve Value in Healthcare.
Brief Title: Scool of Pain (SchooP): A Way to Create Value in Healthcare?
Acronym: SchooP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pernille Friis Rønne, Assistant professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: F-23056260
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Non-cancer Pain; Patient Education as Topic
Keywords: Chronic non-cancer pain; Pain school; Value-based healthcare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain school participants (Experimental)
  Interventions: Other: Pain school intervention

INTERVENTIONS:
Other: Pain school intervention — The pain school intervention consists of seven sessions of two hours duration, varying between teaching, joint reflections, and exercises, carried out once a week for up to 15 patients. The pain school intervention is framed by a biopsychosocial approach, delivered by a team of by multidisciplinary pain specialists. A temporary version of the pain scholl intervention was presented for patient representatives and refined according to their comments.
  The topics of the final pain school sessions include:
  1) Welcome and introduction, 2) Effect and side effects of medication, 3) Balancing demands and resources, 4) Social relationships, 5) Sleep, sofa, and sex, 6) Everyday life, 7) Completion and networking.

SUMMARY:
BACKGROUND: Chronic non-cancer pain (CNCP) is a disabling condition with radical consequences. Magic fix-it solutions do not exist. CNCP is a condition for life, calling for healthcare services supporting its management. Value-based healthcare is a method to work with healthcare that, in the Capital Region of Denmark, serves as a framework for clinicians, administrators, and politicians to deliver healthcare services that create value for patients within available resources. An investigation conducted in collaboration between the Danish Health Association and Danish Regions, involving patients, medical experts, municipality representatives, and general practitioners found that the following preferences should be addressed to achieve value-based healthcare in multidisciplinary treatment of CNCP: Quality of life; acceptance; maintenance, and labor market; communication; social life; sleep; physical status and energy administration; pain management and -relief; emotional status and mood.

In response to the requirement to provide value in healthcare, the Multidisciplinary Pain Centre at Rigshospitalet designed a pain school intervention based on identified preferences. Previous studies have documented the benefits of educational programs in the multidisciplinary treatment of CNCP, but also ethnic/racial and socioeconomic disparities in treatment responses. The present study AIMED to evaluate patients' experience of participating in a pain school, designed to create value in healthcare in the multidisciplinary treatment of CNCP.

DETAILED DESCRIPTION:
DESIGN: The pain school intervention was evaluated using a questionnaire completed by the participants immediately after each of the seven pain school sessions. The questionnaire had two questions: 1: The topic of the pain school session was relevant for me. 2: The teachers communicated the topic of the pain school session appropriately. After the seventh and last pain school session, the participants were also asked to provide an overall evaluation of the pain school using a questionnaire with 9 questions across 4 categories.

The pain school was additionally evaluated using a qualitative design, with focus group interviews with pain school participants and individual interviews with patients who had three or more no-shows or cancellations.

ELIGIBILITY:
The pain school participants were referred to the pain school by the multidisciplinary healthcare provides from the study setting in cohesion with the following criteria:

Inclusion criteria

* Patient motivation
* Ability to join a group and attend a classroom for 2 hours
* Logistical feasibility
* Sufficient energy

Exclusion cireteria

* Inability to understand and speak Danish
* Anxiety
* Depression
* Current resource-demanding opioid-tapering
* Unstable attendance to appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
The topic of the pain school session was relevant for me? | Day 1.
  The Question had five response categories ranging from zero (not at all) to four (to a very great extent).
The teachers communicated the topic of the pain school session appropriately. | Day 1.
  The Question had five response categories ranging from zero (not at all) to four (to a very great extent).

OTHER OUTCOMES:
Overall evaluation of the pain school asking nine questions within four categories. | Day 1.
  Each question item has five respons categories ranging from very dissatisfied to very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Multidisciplinary Paincenter, Department of Anaesthesia, Pain, and Respiratory Support, the Neuroscience Center, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danish Regions. Værdi for patienten, et pejlemærke for fremtidens sundhedsvæsen [Value for the patient - a guiding principle for the future healthcare system]. 2019. https://www.regioner.dk/media/11352/vbspjece-marts19-tryk.pdf
- [Background] The Capital Region of Denmark. Hovedstaden, R. Model for værdibaseret sundhed i Region Hovedstaden [Model for Value-Based Healthcare in the Capital Region of Denmark]. 2020.
- [Background] Porter, ME, & Teisberg, EO. Redefining health care : creating value-based competition on results. Harvard Business School Press, 2006.
- [Background] Huffman KL, Mandell D, Lehmann JK, Jimenez XF, Lapin BR. Clinical and Demographic Predictors of Interdisciplinary Chronic Pain Rehabilitation Program Treatment Response. J Pain. 2019 Dec;20(12):1470-1485. doi: 10.1016/j.jpain.2019.05.014. Epub 2019 Jun 5. PMID 31175957
- [Background] Turner BJ, Liang Y, Rodriguez N, Bobadilla R, Simmonds MJ, Yin Z. Randomized Trial of a Low-Literacy Chronic Pain Self-Management Program: Analysis of Secondary Pain and Psychological Outcome Measures. J Pain. 2018 Dec;19(12):1471-1479. doi: 10.1016/j.jpain.2018.06.010. Epub 2018 Aug 24. PMID 30012494
- [Background] Turner BJ, Rodriguez N, Bobadilla R, Hernandez AE, Yin Z. Chronic Pain Self-Management Program for Low-Income Patients: Themes from a Qualitative Inquiry. Pain Med. 2020 Feb 1;21(2):e1-e8. doi: 10.1093/pm/pny192. PMID 30312459
- [Background] Bruns EB, Befus D, Wismer B, Knight K, Adler SR, Leonoudakis-Watts K, Thompson-Lastad A, Chao MT. Vulnerable Patients' Psychosocial Experiences in a Group-Based, Integrative Pain Management Program. J Altern Complement Med. 2019 Jul;25(7):719-726. doi: 10.1089/acm.2019.0074. PMID 31314560
- [Background] Pate JW, Tran E, Radhakrishnan S, Leaver AM. The Importance of Perceived Relevance: A Qualitative Evaluation of Patient's Perceptions of Value and Impact Following a Low-Intensity Group-Based Pain Management Program. Medicina (Kaunas). 2021 Jan 7;57(1):46. doi: 10.3390/medicina57010046. PMID 33430427
- [Background] Clauw DJ, Essex MN, Pitman V, Jones KD. Reframing chronic pain as a disease, not a symptom: rationale and implications for pain management. Postgrad Med. 2019 Apr;131(3):185-198. doi: 10.1080/00325481.2019.1574403. Epub 2019 Feb 11. PMID 30700198
- [Background] Turk DC, Wilson HD, Cahana A. Treatment of chronic non-cancer pain. Lancet. 2011 Jun 25;377(9784):2226-35. doi: 10.1016/S0140-6736(11)60402-9. PMID 21704872
- [Background] Suso-Ribera C, Yakobov E, Carriere JS, Garcia-Palacios A. The impact of chronic pain on patients and spouses: Consequences on occupational status, distribution of household chores and care-giving burden. Eur J Pain. 2020 Oct;24(9):1730-1740. doi: 10.1002/ejp.1616. Epub 2020 Jul 20. PMID 32533892
- [Background] Caceres-Matos R, Gil-Garcia E, Barrientos-Trigo S, Porcel-Galvez AM, Cabrera-Leon A. Consequences of Chronic Non-Cancer Pain in adulthood. Scoping Review. Rev Saude Publica. 2020 Apr 17;54:39. doi: 10.11606/s1518-8787.2020054001675. eCollection 2020. PMID 32321056
- [Background] Stone AL, Wilson AC. Transmission of risk from parents with chronic pain to offspring: an integrative conceptual model. Pain. 2016 Dec;157(12):2628-2639. doi: 10.1097/j.pain.0000000000000637. PMID 27380502
- [Background] Toye F, Seers K, Hannink E, Barker K. A mega-ethnography of eleven qualitative evidence syntheses exploring the experience of living with chronic non-malignant pain. BMC Med Res Methodol. 2017 Aug 1;17(1):116. doi: 10.1186/s12874-017-0392-7. PMID 28764666
- [Background] Morales-Espinoza EM, Kostov B, Salami DC, Perez ZH, Rosalen AP, Molina JO, Gonzalez-de Paz L, Momblona JMS, Areu JB, Brito-Zeron P, Ramos-Casals M, Siso-Almirall A; CPSGPC Study Group. Complexity, comorbidity, and health care costs associated with chronic widespread pain in primary care. Pain. 2016 Apr;157(4):818-826. doi: 10.1097/j.pain.0000000000000440. PMID 26645546
- [Background] Mills SEE, Nicolson KP, Smith BH. Chronic pain: a review of its epidemiology and associated factors in population-based studies. Br J Anaesth. 2019 Aug;123(2):e273-e283. doi: 10.1016/j.bja.2019.03.023. Epub 2019 May 10. PMID 31079836
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143